CLINICAL TRIAL: NCT00429104
Title: Phase II Study of GM-CSF to Overcome Herceptin-Resistant HER-2/Neu-Overexpressing Metastatic Breast Cancer
Brief Title: Herceptin and GM-CSF for Metastatic Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DM01-0100
Record Dates: First submitted 2007-01-29; First posted 2007-01-31 (Estimated); Results first posted 2011-04-15 (Estimated); Last update posted 2012-12-06 (Estimated); Status verified 2012-12

CONDITIONS: Breast Cancer
Keywords: Breast Cancer; Carcinoma of the Breast; HER-2/neu Overexpression; Herceptin; Trastuzumab; GM-CSF; Sargramostim; Leukine
MeSH Terms: conditions — Breast Neoplasms | interventions — Trastuzumab; Granulocyte-Macrophage Colony-Stimulating Factor; sargramostim

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- HER2+ Metastatic Breast Cancer (Experimental): Herceptin 4 mg/kg IV Over 90 Minutes + GM-CSF 250 mcg/m^2 subcutaneously
  Interventions: Drug: Herceptin; Drug: GM-CSF

INTERVENTIONS:
Drug: Herceptin — 4 mg/kg IV Over 90 Minutes
  Other Names: Trastuzumab
Drug: GM-CSF — 250 mcg/m^2 Subcutaneously
  Other Names: Sargramostim; Leukine

SUMMARY:
Primary Objectives:

1. To determine the patient's tumor response rate that this protocol will produce.
2. To determine the 1 year progression-free survival that this protocol will produce.

Secondary Objective:

1. To determine whether antibody-dependent cell-mediated cytotoxicity (ADCC) is the mechanism of overcoming Herceptin-resistance by use of Granulocyte-Macrophage Colony Stimulating Factor (GM-CSF).

DETAILED DESCRIPTION:
GM-CSF stimulates the immune system and may increase the effectiveness of Herceptin.

Before you can start treatment on this study, you will have what are called "screening tests." These tests will help the doctor decide if you are eligible to take part in this study. You will have a complete medical history and physical exam. This includes blood tests (about 2 tea spoons), and x-rays. Women who are able to have children must have a negative blood or urine pregnancy test.

If you are found to be eligible to take part in this study, you will receive trastuzumab through a vein (IV) every week until the disease gets worse. GM-CSF will be injected under the skin at least once a day until the white blood cell count is stable. GM-CSF will also continue during the course of study until the disease progresses.

You will have further evaluation of your disease by computed tomography-CT scan, bone scan, chest X-ray, etc. at 2, 4, 6, 9, 12, 18, and 24 months after the start of treatment. You will have blood tests (about 2 tea spoons) at least twice a week until the appropriate dose of GM-CSF is found. The dose may increase or decrease depending on the blood test.

You will have blood (about 2 tablespoons) drawn before treatment at the 2nd and 4th month, and if the disease gets worse.

You will be removed from the study if the disease is progressing or severe side effects occur.

This is an investigational study. The FDA has approved trastuzumab and GM-CSF, but their use in this study is experimental. A total of 36 patients will take part in this study. All will be enrolled at UT MD Anderson Cancer Center.

ELIGIBILITY:
Inclusion Criteria:

1. Histological confirmation of invasive carcinoma of the breast.
2. HER-2/neu overexpression: 3+ by immunohistochemical staining or Fluorescence in situ hybridization (FISH) (+).
3. Stage IV breast cancer with measurable disease.
4. Patient receiving progressive disease after Herceptin plus chemotherapy or Herceptin alone. No more than two Herceptin containing regimens.
5. Zubrod performance status 0 or 1.
6. Adequate hematological parameters (White Blood cells-WBC > 3,000/mm3, platelet count > 100,000/mm3), adequate renal function (serum creatinine < 2.0 mg/dl), adequate liver function (total bilirubin, aspartate aminotransferase (AST or SGOT) or alanine aminotransferase (ALT or SGPT) < 3 x normal).

Exclusion Criteria:

1. Active Brain metastasis.
2. No measurable disease at the time of registration (e.g. bone only, leptomeningeal disease alone or pleural effusion alone).
3. More than 2 Herceptin containing regimens in metastatic breast cancer.
4. Known history of HIV positive.
5. Chronic active hepatitis or cirrhosis.
6. Symptomatic pulmonary disease.
7. Use of steroid of non-steroidal anti-inflammatory analgesic or Cox-2 inhibitor 1 week prior to registration.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2002-08; Primary Completion 2009-11 (Actual); Study Completion 2009-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Naoto Ueno, MD, PhD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- U.T.M.D. Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: The University of Texas M.D.Anderson Cancer Center — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment Period of November 2002 to April 2007, all recruited at University of Texas MD Anderson Cancer Center.
Groups:
- HER2+ Metastatic Breast Cancer: Herceptin 4 mg/kg intravenous (IV) Over 90 Minutes + Granulocyte-Macrophage Colony Stimulating Factor (GM-CSF) 250 mcg/m^2 subcutaneously
Period: Overall Study
Arm/Group | HER2+ Metastatic Breast Cancer
Started | 18
Completed | 17
Not Completed | 1
Not completed — Protocol Violation | 1

BASELINE CHARACTERISTICS:
Arm/Group | HER2+ Metastatic Breast Cancer
Number analyzed (Participants) | 18
Age Continuous [Median (Full Range); unit: years] | 48 [27 to 75]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18
  Male | 0
Region of Enrollment [Number; unit: participants]
  United States | 18

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Tumor Response (Stable Disease)
Description: Number of participants with response defined as stable disease or better using Response Evaluation Criteria In Solid Tumors (RECIST) at the month 2 evaluation.
Time Frame: 2 months
Population: Analysis was per protocol, and of 18 enrolled, one participant was inevaluable.
Measure: Number; unit: participants
Arm/Group | HER2+ Metastatic Breast Cancer
Number analyzed (Participants) | 17
participants | 5

2. Secondary Outcome: Duration of Stable Disease
Description: Stable disease is measured from the start of the treatment until the RECIST criteria for disease progression is met.
Time Frame: 6 Years
Population: Analysis was per protocol, and of 18 enrolled, one participant was inevaluable.
Measure: Median (Full Range); unit: weeks
Arm/Group | HER2+ Metastatic Breast Cancer
Number analyzed (Participants) | 17
weeks | 15.8 [10 to 53.9]

ADVERSE EVENTS:
Time Frame: 4 years and 6 months
Arm/Group | HER2+ Metastatic Breast Cancer
Serious Adverse Events (participants affected / at risk) | 0/17
Other Adverse Events (participants affected / at risk) | 17/17
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | HER2+ Metastatic Breast Cancer (N=17)
Fever (Gastrointestinal disorders) | 3
Nausea (Gastrointestinal disorders) | 2
Vomitting (Gastrointestinal disorders) | 1
Sore Mouth (General disorders) | 2
Diarrhea (Gastrointestinal disorders) | 3
Constipation (Gastrointestinal disorders) | 1
Fatigue (General disorders) | 5
Muscle Pain (Musculoskeletal and connective tissue disorders) | 4
Numbness (Nervous system disorders) | 1
Sore finger/toes (Nervous system disorders) | 1
Red eye (Eye disorders) | 1
Rash at injection site (Skin and subcutaneous tissue disorders) | 7
Skin Rash (Skin and subcutaneous tissue disorders) | 6
Itchy hands/feet (General disorders) | 1
Headache (General disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No